CLINICAL TRIAL: NCT05061069
Title: Implementation of a Standard Vestibular Screening Protocol for Hearing-impaired Infants in Flanders
Brief Title: Vestibular Infants Screening-Flanders
Acronym: VIS-Flanders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: Universitair Ziekenhuis Brussel (Other); Universitaire Ziekenhuizen KU Leuven (Other); Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other); Queen Fabiola Children's University Hospital (Other); AZ Turnhout (Other); Gasthuis Zusters Antwerpen (Other); GZA Ziekenhuizen Campus Sint-Augustinus (Other); University Hospital, Antwerp (Other); Jessa Hospital (Other); Ziekenhuis Oost-Limburg (Other); Algemeen Stedelijk Ziekenhuis (Other); Algemeen Ziekenhuis Maria Middelares (Other); AZ Delta (Other); AZ Sint-Jan AV (Other); AZ Sint-Lucas Brugge (Other); Sint-Lievenspoort Gent (Unknown); Center for Developmental and Hearing Disorders (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2018/0435 (BC-2604); T000917N (Other Grant/Funding Number: Research Foundation-Flanders)
Record Dates: First submitted 2021-09-09; First posted 2021-09-29 (Actual); Results first posted 2025-02-12 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-01

CONDITIONS: Vestibular Disorder; Hearing Impaired Children
Keywords: vestibular; balance; hearing loss; infants
MeSH Terms: conditions — Vestibular Diseases; Hearing Loss | interventions — Vestibular Evoked Myogenic Potentials

STUDY DESIGN:
Intervention Model Description: Multicenter non-commercial interventional academic research
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Infants with permanent hearing loss (Experimental): Each infant with permanent hearing loss in Flanders will be offered a vestibular screening by means of the cVEMP (cervical vestibular evoked myogenic potentials) test to screen for vestibular deficits.
  Interventions: Diagnostic Test: cervical vestibular evoked myogenic potentials (cVEMP)

INTERVENTIONS:
Diagnostic Test: cervical vestibular evoked myogenic potentials (cVEMP) — cVEMPs are ipsilateral, short latency, inhibitory myogenic potentials that assess otolith (mainly saccular) function and the integrity of the inferior branch of the vestibular nerve.

SUMMARY:
Hearing-impaired children are at risk for a vestibular impairment, as the auditory and vestibular end organs are closely related. Although this can compromise a child's development on many levels, vestibular testing is not routinely performed in this vulnerable group. This project aims to give each congenitally hearing-impaired child in Flanders (Belgium) access to a basic vestibular screening at a young age and set an example for other regions worldwide.

DETAILED DESCRIPTION:
The implementation of a vestibular screening in hearing-impaired babies of six months old will timely discover vestibular problems to limit the impact on the (motor) development. The cervical vestibular evoked myogenic potential (cVEMP) technique will be used as a vestibular screening tool. Flanders is the first region worldwide that will implement a vestibular screening. All official Flemish reference centres of Kind en Gezin (Child and Family) will participate in this project.

Study purpose:

The final utilisation goal of this project is to limit the impact of a vestibular dysfunction on the (motor) development of children. Since hearing-impaired children have a higher risk for deficits of the vestibular (balance) organ, the researchers will focus on this vulnerable group.

This will be accomplished by:

* The implementation of a standard vestibular screening protocol in Flanders in hearing-impaired children at the age of 6 months, enabling early diagnosis of vestibular deficits and adequate referral for extensive vestibular testing, motor assessment and rehabilitation.
* Increasing the awareness for vestibular dysfunctions and its associated symptoms in hearing-impaired children among parents, teachers, paramedics, specialists and other social workers who are in close contact with hearing-impaired children. This should go hand in hand with more effective patient care, because adequate therapy will start sooner.

Methodology:

The aim of the project is to add a vestibular screening to the existing auditory screening programme (MAICO test). The following steps will be performed to guarantee an accurate vestibular follow-up in Flemish hearing-impaired children:

* In case of a 'refer' on the second MAICO test, Kind en Gezin (Child and Family) will refer the child to the reference centres of Kind en Gezin in Flanders.
* These reference centres will perform a diagnostic hearing test (brainstem evoked response audiometry: BERA) to confirm the permanent hearing loss (standard of care).
* Each child with a confirmed hearing loss (BERA 'refer') will be subjected to a vestibular screening at the age of six months (on average 120/year), combined with tympanometry, in that specific reference centre at the age of six months. The cervical vestibular evoked myogenic potential (cVEMP) technique will be used.
* In case of a refer on the vestibular screening (cVEMP 'refer'), the reference centres will refer the child for motor assessment and, if necessary, for rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Flemish children with permanent congenital or delayed-onset hearing loss, which occurred before the age of 9 months, are included.

Exclusion Criteria:

* Children with temporary hearing loss (e.g. due to otitis media) are excluded.

Ages: 4 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 301 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2022-08-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leen Maes, Prof. Dr., Study Director — University Ghent; Ingeborg Dhooge, Prof. Dr., Principal Investigator — University Hospital, Ghent
Locations (19):
- Belgium (19):
  - Ghent University Hospital, Ghent, East-Flanders
  - Algemeen Stedelijk Ziekenhuis, Aalst
  - Algemeen Ziekenhuis Maria Middelares, Aalst
  - Eargroup, Antwerp
  - Gasthuis Zusters Antwerpen, Antwerp
  - GZA Ziekenhuizen Campus Sint-Augustinus, Antwerp
  - University Hospital Antwerp, Antwerp
  - AZ Sint-Jan, Bruges
  - AZ Sint-Lucas Brugge, Bruges
  - Cliniques universitaires Saint-Luc, Brussels
  - Queen Fabiola Children's University Hospital, Brussels
  - Universitair Ziekenhuis Brussel, Brussels
  - Ziekenhuis Oost-Limburg, Genk
  - Sint-Lievenspoort Gent, Ghent
  - Jessa Hospital, Hasselt
  - Universitair Ziekenhuis Leuven, Leuven
  - AZ Delta, Menen
  - CAR Stappie, Ostend
  - AZ Turnhout, Turnhout

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared as data related to health of patients is included.

REFERENCES:
- [Background] Martens S, Dhooge I, Dhondt C, Leyssens L, Sucaet M, Vanaudenaerde S, Rombaut L, Maes L. Vestibular Infant Screening - Flanders: The implementation of a standard vestibular screening protocol for hearing-impaired children in Flanders. Int J Pediatr Otorhinolaryngol. 2019 May;120:196-201. doi: 10.1016/j.ijporl.2019.02.033. Epub 2019 Feb 25. PMID 30849604
- [Result] Martens S, Dhooge I, Dhondt C, Vanaudenaerde S, Sucaet M, Rombaut L, Boudewyns A, Desloovere C, Janssens de Varebeke S, Vinck AS, Vanspauwen R, Verschueren D, Foulon I, Staelens C, Van den Broeck K, De Valck C, Deggouj N, Lemkens N, Haverbeke L, De Bock M, Oz O, Declau F, Devroede B, Verhoye C, Maes L. Vestibular Infant Screening (VIS)-Flanders: results after 1.5 years of vestibular screening in hearing-impaired children. Sci Rep. 2020 Dec 3;10(1):21011. doi: 10.1038/s41598-020-78049-z. PMID 33273502
- [Result] Dhondt C, Maes L, Rombaut L, Martens S, Vanaudenaerde S, Van Hoecke H, De Leenheer E, Dhooge I. Vestibular Function in Children With a Congenital Cytomegalovirus Infection: 3 Years of Follow-Up. Ear Hear. 2021 Jan/Feb;42(1):76-86. doi: 10.1097/AUD.0000000000000904. PMID 32590628
- [Derived] Martens S, Dhooge I, Dhondt C, Vanaudenaerde S, Sucaet M, Van Hoecke H, De Leenheer E, Rombaut L, Boudewyns A, Desloovere C, Vinck AS, de Varebeke SJ, Verschueren D, Verstreken M, Foulon I, Staelens C, De Valck C, Calcoen R, Lemkens N, Oz O, De Bock M, Haverbeke L, Verhoye C, Declau F, Devroede B, Forton G, Deggouj N, Maes L. Three Years of Vestibular Infant Screening in Infants With Sensorineural Hearing Loss. Pediatrics. 2022 Jul 1;150(1):e2021055340. doi: 10.1542/peds.2021-055340. PMID 35698886
- See also: VIS-Flanders website for patients and health care workers — http://VIS-Flanders.be/en/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The vestibular screening was offered to all Flemish infants with permanent hearing loss around the age of 6 months in 1 of the 25 reference centers involved in the UNHSP.
Period: Overall Study
Arm/Group | Infants With Permanent Hearing Loss
Started | 301
Completed | 301
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 301 infants were screened, 47 were excluded for analysis, so the cVEMP data of 254 infants was eventually included and analyzed.
Arm/Group | Infants With Permanent Hearing Loss
Number analyzed (Participants) | 301
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 301
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: months] | 7.4 (2.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 153
  Male | 148
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Belgium | 301
Infant with permanent hearing loss [Count of Participants; unit: Participants] | 301

OUTCOME MEASURES:

1. Primary Outcome: Number of Hearing-impaired Infants in Flanders With Abnormal Vestibular Screening Results.
Description: The primary outcome measure is the number of hearing-impaired infants in Flanders with abnormal vestibular screening results according to the degree, laterality, and onset of hearing loss. Abnormality of the vestibular screening results is based on the rectified interpeak amplitude values of the cVEMP (cervical vestibular evoked myogenic potentials) responses.
Time Frame: Each infants will be subjected to the screening at the age of six months. In case of inconclusive results during the first screening, the screening will be repeated within three months after the first screening moment.
Population: Overall, 301 infants were screened, of which 47 infants were excluded for data analysis.
  Excluded infants:
  Bilateral normal hearing during audiological follow-up: n = 9 Parents declined retest in case of initial inconclusive results: n = 6 Delayed-onset hearing loss after ten months of age: n = 1 Permanent conductive hearing loss due to external auditory canal atresia: n = 22 Parents gave consent to perform the cVEMP, but did not give consent to analyze and include the data: n = 9
Measure: Count of Participants; unit: Participants
Arm/Group | Infants With Permanent Hearing Loss
Number analyzed (Participants) | 254
Participants | 35

ADVERSE EVENTS:
Description: All-cause mortality, serious, and other (not including serious) adverse events were not monitored/assessed.
Arm/Group | Infants With Permanent Hearing Loss
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-05-21): https://cdn.clinicaltrials.gov/large-docs/69/NCT05061069/Prot_SAP_000.pdf